CLINICAL TRIAL: NCT01248052
Title: Single-Ascending Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of LY2979165 in Healthy Subjects
Brief Title: A First Human Dose Study to Investigate Safety and Tolerability of LY2979165 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13844; I4S-EW-HHCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY2979165 (Part A) (Experimental): single oral doses at dose levels ranging from 20 to 1000 mg
  Interventions: Drug: LY2979165
- Placebo (Part A) (Placebo Comparator): single oral dose
  Interventions: Drug: Placebo
- LY2979165 - low dose (Part B) (Experimental): single oral low dose of LY297165 (dose to be determined by Part A)
  Interventions: Drug: LY2979165
- LY2979165 - high dose (Part B) (Experimental): single oral high dose of LY2979165 (dose determined from Part A)
  Interventions: Drug: LY2979165
- Placebo - Part B (Placebo Comparator): single oral dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2979165 — administered orally
  Arms: LY2979165 (Part A); LY2979165 - high dose (Part B); LY2979165 - low dose (Part B)
Drug: Placebo — administered orally
  Arms: Placebo (Part A); Placebo - Part B

SUMMARY:
This is a two part study (Parts A and B), the purpose of which is to determine the safety of LY2979165 in healthy people, and any side effects that might be associated with it, and to understand how the body handles LY2979165. In addition, Part B, will also look at levels of LY2979165 in spinal fluid. Doses investigated will be in the range of 20-1000 mg.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination. Female subjects in Part B are at the site's discretion.
* Male subjects: Agree to use a reliable method of birth control during the study.
* Female subjects: Women not of child-bearing potential due to surgical sterilisation (hysterectomy or bilateral oophorectomy or tubal ligation) or postmenopausal as defined by age greater than or equal to 45 years with an intact uterus, who have not taken hormones or oral contraceptives for > 1 year, and either:

  * spontaneous amenorrhea of >12 months, or
  * spontaneous amenorrhea of 6-12 months with a follicle- stimulating hormone (FSH) level of >40 mIU/mL
* Are between the body mass index (BMI) of 18.5 and 29.9 kg/m2, inclusive.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the ethical review board governing the site.

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device, other than the study drug/device used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Are persons who have previously completed or withdrawn from this study.
* History of clinically significant adverse drug reactions or "drug allergy" to more than 3 different types of systemically administered medications or known allergies to LY2979165 or it's constituents.
* Have a Bazett's corrected QT (QTcB) interval value of >450 msec (males) or >470 msec (females) or any abnormality in the screening 12-lead ECG that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Have an abnormal blood pressure (at least 5 minutes in supine position) as determined by the investigator.
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, immunological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have increased risk of seizures as evidenced by a history of: greater than or equal to 1 seizure (except childhood febrile seizure), history of electroencephalogram with epileptiform activity, history of stroke, surgery to the cerebral cortex, or head trauma with loss of consciousness.
* Show evidence of significant active neuropsychiatric disease.
* Have a history of alcohol or drug abuse.
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen.
* Have donated blood of more than 450 mL within the last 3 months prior to dosing.
* Intended use of over-the-counter medication within 7 days prior to dosing or during the study with the exception of vitamins and mineral supplements (not providing >100% of the recommended dietary allowance [RDA]), or occasional paracetamol or acetaminophen. If this situation arises, inclusion of an otherwise suitable subject may be at the discretion of the sponsor.
* Intended use of herbal supplements or prescription medications, other than stable doses of thyroid or estrogen hormone replacement, within 14 days prior to dosing or during the study. If this situation arises, inclusion of an otherwise suitable subject may be at the discretion of the sponsor.
* Subjects who meet at least 1 of the following criteria (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits):

  * subjects who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females),
  * subjects unwilling to stop alcohol consumption 48 hours prior to dosing until the completion of each study appointment, or
  * subjects unwilling to limit alcohol intake to no more than 3 units per day between study appointments.
* Cigarette consumption of more than 10 cigarettes per day or unable/unwilling to abide by CRU smoking restrictions during admissions.
* Any other condition, which in the opinion of the investigator, would preclude participation in the study.

In addition for Part B only:

* Abnormalities in lumbar spine previously known or determined by screening lumbar x-ray.
* History of clinically significant back pain, back pathology and/or back injury (for example, degenerative disease, spinal deformity or spinal surgery) that may predispose to complications or technical difficulty with lumbar puncture.
* Have evidence or history of significant active bleeding or coagulation disorder or have taken non-steroidal anti inflammatory drugs (NSAIDs) or other drugs that affect coagulation or platelet function within 14 days prior to lumbar catheter insertion.
* Have an allergy to lidocaine (Xylocaine®) or its derivatives.
* Have medical or surgical conditions in which lumbar puncture is contraindicated.
* Have participated in Part A of this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant effects | predose through 48 hours postdose

SECONDARY OUTCOMES:
Pharmacokinetics, area under the concentration curve (AUC), Parts A and B | predose through 48 hours postdose
Pharmacokinetics maximum plasma concentration (Cmax), Parts A and B. | predose through 48 hours post dose
Pharmacokinetics, cerebrospinal fluid area under the concentration curve (AUC), Part B only | predose through 48 hours postdose
Pharmacokinetics, maximum cerebrospinal fluid concentration (Cmax), Part B only | predose through 48 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Singapore, Singapore